CLINICAL TRIAL: NCT06383455
Title: Effects of Smoking on Clinical and Microbiological Response Following Non-Surgical Periodontal Treatment in Periodontitis Patients
Brief Title: Effects of Smoking on Clinical and Microbiological Response in Individuals With Periodontitis
Status: Completed | Type: Observational
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Ece AÇIKGÖZ ALPARSLAN, Assisstant Professor, Trakya University
Other Study IDs: Observational
Record Dates: First submitted 2024-04-18; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Periodontitis; Smoking Habit; Subgingival Plaque
MeSH Terms: conditions — Periodontitis; Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Subgingival microbial dental plaque samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Smoking individuals with periodontitis: The participants were divided into two groups according to self-reported smoking habits. The smoker group consisted of individuals with stage 3/4 periodontitis who smoked at least ten cigarettes per day for at least five years.
  Interventions: Procedure: Non-surgical periodontal therapy
- Non-smoking individuals with periodontitis: The non-smoker group consisted of individuals with Stage 3/4 periodontitis who had never smoked in a lifetime or had quit smoking at least two years ago.
  Interventions: Procedure: Non-surgical periodontal therapy

INTERVENTIONS:
Procedure: Non-surgical periodontal therapy — An ultrasonic device (Cavitron Plus, Dentsply®, Duisburg, Germany) and periodontal hand instruments (periodontal curettes; Chicago, IL) were used for non-surgical periodontal treatment. The treatment procedure also included detailed oral hygiene instructions and full-mouth scaling and root planing. Scaling and root planing (SRP) was applied to all four quadrants under local anesthesia in a single appointment. No medication or mouthwash was prescribed to the patients.

SUMMARY:
This study aimed to compare the distribution of subgingival periodontal pathogens following non-surgical periodontal therapy in smoking and non-smoking people with periodontitis. The main question it aims to answer is:

- Does smoking affect the results of non-surgical periodontal treatment on subgingival flora in participants with periodontal disease?

Researchers performed non-surgical periodontal therapy on 48 participants with stage III/IV periodontitis and recorded clinical measurements. They obtained subgingival plaque samples from periodontal pockets at the onset and after four weeks of treatment, determining the level of periodontopathogens using a polymerase chain reaction-based method.

DETAILED DESCRIPTION:
The present study aims to compare the changes in clinical parameters and subgingival periodontopathogen rates (P. gingivalis, A. actinomycetemcomitans, T. forsythia, F. nucleatum, P. intermedia, T. denticola, P. micra, C. rectus, E. nodatum, Capnocytophaga spp, and E. corrodens) following full-mouth scaling and root planing procedures in participants with and without smoking habits.

ELIGIBILITY:
Inclusion Criteria:

* Having 15 or more permanent teeth (except third molars and teeth with endodontic lesions),
* Having been diagnosed with generalized Stage III or IV periodontitis that progresses with periodontal support tissue loss in more than 30% of the teeth,
* Having at least five teeth with probing depth(PD) ≥6mm, clinical attachment level(CAL) ≥5mm, and radiographic bone loss that extends to at least the middle of the root,
* Having at least one tooth that meets the same PD and CAL criteria per quadrant.

Exclusion Criteria:

* Pregnancy or lactation,
* Any systemic disease with a potential influence on the immune response (diabetes mellitus, bone metabolic diseases, immunosuppressive therapy, radiation etc.),
* Existence of decay, restoration, or prosthesis on the sampling site,
* Use of the anti-inflammatory drug and antibiotic within the last 3 months.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consisted of a total of 48 systemically healthy adults who applied to the Trakya University Faculty of Dentistry with periodontal complaints. The participants had generalized stage III/IV periodontitis, determined according to the criteria stated by the 2017 World Workshop for the Classification of Periodontal Diseases and Conditions. These participants were divided into two groups according to self-reported smoking habits.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Change in levels of periodontopathogens in subgingival plaque after non-surgical periodontal therapy in smokers and non-smokers with stage 3/4 periodontitis | Baseline and four weeks after the periodontal therapy.
  The baseline levels of periodontopathogens (P. gingivalis, A. actinomycetemcomitans, T. forsythia, F. nucleatum, P. intermedia, T. denticola, P. micra, C. rectus, E. nodatum, Capnocytophaga spp, and E. corrodens), post-treatment levels, and elimination levels with treatment were evaluated using multiplex polymerase chain reaction (PCR) analysis.The observed rates of microorganisms were assessed by determining six main levels.
  0: No colouring (<1% no bacteria)
  1. Very light-colored staining (Determination of bacteria from 1% to 20%).
  2. Light colored staining (Determination of bacteria from 21% to 40%),
  3. Moderate colored staining (Determination of bacteria from 41% to 60%),
  4. Dark colored staining (Determination of bacteria from 61% to 80%),
  5. Very dark-colored staining (Determination of bacteria from 81% to 100%).

SECONDARY OUTCOMES:
Change in clinical attachment level (CAL) | Baseline and 4 weeks after periodontal therapy
  CAL is the main clinical parameter indicating the severity of periodontal disease. CAL measurements were performed on six different surfaces of each tooth (disto-buccal/labial, mid-buccal/labial, mesio-buccal/labial, disto-lingual, mid-lingual, and mesio lingual) by using a periodontal probe (Williams probe; Chicago, IL) and average value was calculated in millimeters.
  CAL 1-2 mm: Stage 1 periodontitis CAL 3-4 mm: Stage 2 periodontitis CAL ≥ 5 mm: Stage 3/4 periodontitis
Change in probing depth (PD) | Baseline and 4 weeks after periodontal therapy
  PD is one of the clinical parameters indicating the severity of periodontal disease. PD measurements were performed on six different surfaces of each tooth (disto-buccal/labial, mid-buccal/labial, mesio-buccal/labial, disto-lingual, mid-lingual, and mesio lingual) by using a periodontal probe (Williams probe; Chicago, IL) and average value was calculated in millimeters.
  PD ≤ 4 mm: Stage 1 periodontitis PD ≤ 5 mm: Stage 2 periodontitis PD ≥ 6 mm: Stage 3/4 periodontitis
Change in gingival index (GI) scores | Baseline and 4 weeks after periodontal therapy
  GI is a clinical parameter indicating the severity of gingival inflammation. GI scores were noted for four different surfaces of each tooth (buccal, distal, mesial and lingual) and average value was calculated.
  0 = normal gingiva;
  1. = mild inflammation: slight change in color, slight edema, no bleeding on probing;
  2. = moderate inflammation: redness, edema, and glazing, or bleeding on probing;
  3. = severe inflammation: marked redness and edema, tendency toward spontaneous bleeding.
Change in plaque index (PI) scores | Baseline and 4 weeks after periodontal therapy
  PI is a clinical parameter indicating the severity of dental plaque accumulation and oral hygiene habits of individuals. PI scores were noted for four different surfaces of each tooth (buccal, distal, mesial and lingual) and average value was calculated.
  0 = No plaque
  1. = A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or by using the probe on the tooth surface.
  2. = Moderate accumulation of soft deposits within the gingival pocket, or the tooth and gingival margin which can be seen with the naked eye.
  3. = Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
Change in Bleeding on Probing (BOP) | Baseline and 4 weeks after periodontal therapy
  BOP is one the clinical parameters indicating the severity of gingival inflammation. BOP were noted as positive or negative for four different surfaces of each tooth (buccal, distal, mesial and lingual) and average positive value was calculated in %.

CONTACTS AND LOCATIONS:
Overall Officials: Ece Açıkgöz-Alparslan, Principal Investigator — Trakya University
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Researchers will consider sharing the entire protocol and statistical plan with other researchers after this study is published as a scientific article

REFERENCES:
- [Background] Kubota M, Tanno-Nakanishi M, Yamada S, Okuda K, Ishihara K. Effect of smoking on subgingival microflora of patients with periodontitis in Japan. BMC Oral Health. 2011 Jan 5;11:1. doi: 10.1186/1472-6831-11-1. PMID 21208407
- [Background] Van der Velden U, Varoufaki A, Hutter JW, Xu L, Timmerman MF, Van Winkelhoff AJ, Loos BG. Effect of smoking and periodontal treatment on the subgingival microflora. J Clin Periodontol. 2003 Jul;30(7):603-10. doi: 10.1034/j.1600-051x.2003.00080.x. PMID 12834497
- [Background] Labriola A, Needleman I, Moles DR. Systematic review of the effect of smoking on nonsurgical periodontal therapy. Periodontol 2000. 2005;37:124-37. doi: 10.1111/j.1600-0757.2004.03793.x. No abstract available. PMID 15655029
- [Background] Grossi SG, Zambon J, Machtei EE, Schifferle R, Andreana S, Genco RJ, Cummins D, Harrap G. Effects of smoking and smoking cessation on healing after mechanical periodontal therapy. J Am Dent Assoc. 1997 May;128(5):599-607. doi: 10.14219/jada.archive.1997.0259. PMID 9150643
- [Background] Darby IB, Hodge PJ, Riggio MP, Kinane DF. Clinical and microbiological effect of scaling and root planing in smoker and non-smoker chronic and aggressive periodontitis patients. J Clin Periodontol. 2005 Feb;32(2):200-6. doi: 10.1111/j.1600-051X.2005.00644.x. PMID 15691352
- [Background] Haffajee AD, Yaskell T, Torresyap G, Teles R, Socransky SS. Comparison between polymerase chain reaction-based and checkerboard DNA hybridization techniques for microbial assessment of subgingival plaque samples. J Clin Periodontol. 2009 Aug;36(8):642-9. doi: 10.1111/j.1600-051X.2009.01434.x. Epub 2009 Jun 26. PMID 19563330
- [Derived] Acikgoz-Alparslan E, Eryildiz C, Inanc B. Effects of Smoking on Clinical and Microbiological Response Following Non-Surgical Periodontal Treatment in Periodontitis Patients. Int J Dent Hyg. 2025 Nov 25. doi: 10.1111/idh.70007. Online ahead of print. PMID 41290565